CLINICAL TRIAL: NCT04403373
Title: Effectiveness of Different Intensities Walking Exercise in Improving Depression in Older Adults With Major Depressive Disorder, A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Walking Exercise in Improving Depression in Older Adults With Major Depressive Disorder, A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor & Head of Division of Kinesiology, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-9835-MDD-007
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD, Walking Exercise, Exercise Intensity
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded from the group allocation and the participants are instructed not to reveal what kind of intervention he/she received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waitlist control group (Placebo Comparator): Participants in this group receive no intervention during the 12-week period.
  Interventions: Behavioral: Waitlist control
- Moderate-intensity walking group (Experimental): Participants in this group will perform a thrice-a-week walking exercise at a moderate intensity (~3.5 METs). The training will be conducted outdoors. Each training session lasts for 50 minutes.
  Interventions: Behavioral: Moderate-intensity walking exercise
- Vigorous-intensity walking group (Experimental): Participants in this group will perform a thrice-a-week walking exercise at a vigorous intensity (~7 METs). The training will be conducted outdoors. Each training session lasts for 25 minutes.
  Interventions: Behavioral: Vigorous-intensity walking exercise

INTERVENTIONS:
Behavioral: Waitlist control — waitlist control
  Arms: Waitlist control group
Behavioral: Moderate-intensity walking exercise — walking exercise
  Arms: Moderate-intensity walking group
Behavioral: Vigorous-intensity walking exercise — walking exercise
  Arms: Vigorous-intensity walking group

SUMMARY:
1. This pilot randomized controlled trial aims at investigating the effects of different intensities of aerobic walking exercise to alleviate depression in older adults with major depressive disorder. Both baseline and post-intervention measurements will be conducted at the Exercise Physiology Laboratory, Division of Kinesiology, School of Public Health, The University of Hong Kong, while the exercise intervention will be conducted outdoors in a small group setting (3-5 participants).
2. Three-time-per-week moderate-intensity (~3.5 METs) or vigorous-intensity (~7 METs) walking exercise will be prescribed to participants in two exercise groups, while the participants in the waitlist group will receive no intervention. The intervention duration is 12 weeks.
3. We will recruit participants from the community in HK. Interested participants will be invited for a semi-structured interview including an assessment on the Beck Depression Inventory and medical history record to confirm eligibility.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged equal or over 50 years;
2. Ethnic Chinese;
3. Beck Depression Inventory score over 9 points;
4. Diagnosed with MDD and currently on pharmacological treatment for MDD.

Exclusion Criteria:

1. Incapable of participating in physical exercise with major confounding conditions which are known to affect mobility;
2. Cannot walk without assistive device;
3. Regular exercise habit (defined as exercise > 3 times per week and each time > 50 minutes)
4. Any serious somatic condition that prevents walking exercise participation (such as limb loss)
5. History of major diseases e.g. cancer, cardio-/cerebrovascular, neurodegenerative and renal diseases;
6. Diagnosis of dementia/Alzheimer's disease, or currently using antidementia medication;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms-Beck Depression Inventory (BDI) | 3 Months
  BDI is a 21-item self-reporting questionnaire for evaluation of the severity of depression in both normal and psychiatric populations. Each item includes four statements numbered from 0 to 3, with a higher number indicating more severe depressive symptoms. Participants will be asked to circle the statement that can best describe them in a paper-pencil based manner. The BDI score interpretation is: less than 10: no or minimal depression, 10-18: mild-to-moderate depression, 19-29: moderate-to-severe depression, over 30: severe depression

SECONDARY OUTCOMES:
Antidepressants Usage-Medication History | 3 Months
  The use of antidepressants such as most commonly prescribed Prozac (fluoxetine), Zoloft (sertraline), Lexapro (escitalopram), Paxil (paroxetine), Celexa (citalopram), or selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, with detailed usage information (e.g., drug name, type, dosage, and frequency of dosage) will be recorded. Subjects will be asked to provide the dosage, frequency of the daily antidepressant usage. The duration between the first interview of this study and the first diagnosis of MDD will also be recorded.
Anxiety-Generalized Anxiety Disorder 7-item (GAD-7) scale | 3 Months
  Generalized Anxiety Disorder 7-item (GAD-7) scale will be used to measure the anxiety level of the subjects. The GAD-7 is a reliable and valid measure of anxiety severity and its brevity make the GAD-7 a useful clinical and research tool. Higher score indicates more severe level of anxiety.
Sleep quality-Pittsburgh Sleep Quality Index (PSQI) | 3 Months
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized instrument to estimate sleep quantity and quality. The PSQI has been commonly used to distinguish people with primary insomnia from normal sleepers. The Chinese version of PSQI has been validated to have a satisfactory Cronbach's alpha of 0.82-0.83 and test-retest reliability of 0.85 among Hong Kong Chinese older adults.
Quality of life-12-item short form health survey (SF-12) | 3 Months
  SF-12 was originally developed for medical outcomes study, and it is one of the most widely used instruments for assessing health-related quality of life. SF-12 covers the same eight domains as the SF-36 form, which assesses physical functioning, emotional and mental health, body pain, general health, social functioning and vitality, with a higher score indicating a better quality of life.
Cardiorespiratory fitness-VO2max Test | 3 Months
  The participant's maximal oxygen consumption will be measured at baseline, 12 weeks intervention to evaluate the participants' cardiovascular fitness by VO2max test using a COSMED Quark Series telemetric gas analysis system.
Resting heart rate | 3 Months
  The participant will be asked to sit quietly for 20 minutes for resting HR recording. The resting HR will be measured by Optical heart rate sensor (Polar OH1).
Body Mass Index | 3 Months
  Body weight and height of the subject will be measured by a validated scale (A&D, UC-321) to the nearest 0.1kg and stadiometer (SECA, CE-0123) to the nearest 0.1cm. The BMI will be calculated as BMI = kg/m2.
Daily physical activity-International Physical Activity Questionnaire (IPAQ) | 3 Months
  The Chinese version of IPAQ is one of the most reliable self-report measures of physical activity for older adults, with intraclass correlation coefficients ranging from 0.81 to 0.89. Three categories of physical activities are classified in IPAQ: Low, moderate and high. Continuous score is also suggested to be expressed as MET-min per week, which can be calculated using the data from IPAQ.

CONTACTS AND LOCATIONS:
Overall Officials: MING FAI P SIU, Ph.D, Principal Investigator — The University of Hong Kong
Locations (1):
- Li Kai Shing Faculty of Medicine, Hong Kong, Southern District, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.

REFERENCES:
- [Derived] Yu DJ, Yu AP, Leung CK, Chin EC, Fong DY, Cheng CP, Yau SY, Siu PM. Comparison of moderate and vigorous walking exercise on reducing depression in middle-aged and older adults: A pilot randomized controlled trial. Eur J Sport Sci. 2023 Jun;23(6):1018-1027. doi: 10.1080/17461391.2022.2079424. Epub 2022 Jun 13. PMID 35579606